CLINICAL TRIAL: NCT04986449
Title: Nutritional and Culinary Habits to Empower Families (n-CHEF) - A Feasibility Study
Brief Title: Nutritional and Culinary Habits to Empower Families - A Feasibility Study
Acronym: n-CHEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021.036
Record Dates: First submitted 2021-06-25; First posted 2021-08-02 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Family Research
Keywords: culinary medicine; home cooking; feasibility study

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): All families will receive the culinary and nutritional intervention. Changes before-after will be assessed regarding culinary skills, knowledge and attitudes of families on cooking with plant-based foods
  Interventions: Behavioral: nutritional and culinary intervention

INTERVENTIONS:
Behavioral: nutritional and culinary intervention — Each family will attend a total of 4 culinary-nutritional workshops between April and June 2021. Workshops 1 and 2 will be held in the kitchen located at the Science Building of the University of Navarra and will be given individually to each family.
  Workshops 3 and 4 will be online (Zoom) and will be held in groups of 5 families. These workshops will be held from 5.30 pm to 7.30 pm on Fridays or from 11.30 am to 1.30 pm on Saturdays.
  Finally, a meeting will be organized with all the families (parents and children) where the recipes prepared by the children for the n-CHEF challenge will be shared and prizes will be awarded.

SUMMARY:
Background: Currently, one of the health challenges in the field of public health is to improve the quality of life of people with metabolic diseases, using new strategies to promote eating habits and lifestyle that allow an active involvement in health.

Within the new strategies to promote an improvement in the eating habits of the population, culinary-nutritional interventions based on culinary medicine or strategies such as home-cooking, have been proposed as effective measures for the implementation of healthy eating habits in the population. Intervention with families (the environment in which the eating habits of children are implemented for the future) should be highlighted.

Methods: The present project will cover culinary medicine and home-cooking as innovative strategies to improve the eating habits of families through an intervention based on face-to-face (2) and online (2) cooking workshops, where apart from receiving nutritional education, they will be taught a series of culinary techniques (adapted to adults and children) so that they learn to cook in an easy, enjoyable and family-friendly way, with tools to eat healthier in a simple and quick way.

The main objective is to evaluate the feasibility of the culinary-nutritional intervention. The intervention will be carried out with 15 families (one of the parents and one of the children of the family aged between 10 and 14 years), through the measurement of anthropometric parameters and questionnaires on eating habits and lifestyles (both individual and family). In addition, questionnaires specific to the research will be collected in order to study the feasibility of the intervention.

ELIGIBILITY:
The study population is 15 families. The main inclusion criterion is that in the family there is a minor between 10 and 14 years of age. As this is a feasibility study, children will be healthy, although they may be overweight, but not following any special diet.

Inclusion criteria :

* Families in which at least one parent commits to attend all information-gathering visits and culinary-nutritional workshops.
* Families in which the child who commits to attend the information gathering visits and culinary-nutritional workshops is between 10 and 14 years old.
* Families in which the parent and the child eat food prepared at home at least 5 days a week.
* Families that assume the cost of food purchases for the workshops.

Exclusion criteria:

* Families in which children and/or parents eat 5 days a week food not prepared at home.
* Families in which any member of the family has allergies (nuts, fruits, cow protein...) or food intolerances (dairy, gluten...) that prevent them from following the culinary-nutritional intervention.
* Families that follow a specific dietary pattern that makes the intervention impossible (weight loss diet, vegetarian or vegan diet, etc.).
* Families in which some members have chronic diseases such as type 1 diabetes, morbid obesity, type 2 diabetes, etc.
* Families in which one of the parents is involved in cooking and/or nutrition or one of the parents and/or children have attended a previous cooking course.
* Families in which any member has eating disorders (bulimia, anorexia nervosa).
* Families in which any member has severe digestive tract diseases, kidney disease, cancer, and other diseases that limit survival to 1 year.
* Families in which a member presents some type of cognitive and/or psychic impairment, Alzheimer's disease, depressive pathology, etc.
* Families in which poor collaboration is foreseen or that, in the opinion of the researcher, any of the members have difficulties in following the study procedures.
* Families in which a lack of commitment (in the researcher's opinion) to the intervention, suspicion of non-compliance, or real difficulties in following the development of the study are detected.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Effect of the culinary intervention on home cooking habits measured with the Culinary Habits Frequency Questionnaire | 8 months
  A validated questionnaire will be used to assess the use of different culinary techniques (Culinary Habits Frequency Questionnaire). This questionnaire collects information about the frequency use of cooking techniques applied when cooking several food groups during the past year. Answers include 8 different categories, from never to 3 or more times per day. Results between the baseline and 8-month questionnaires will be compared.
Adherence to the Mediterranean Diet (MedDiet) | 8 months
  Adherence to the MedDiet will be measured with a validated 14-item Mediterranean Diet Adherence (MEDAS) questionnaire. A higher score means a higher adherence to the Mediterranean Diet. Results between the baseline and 8-month questionnaires will be compared.
Home cooking attitudes and self-confidence on cooking at home with the cooking attitudes and self-confidence questionnaire | 8 months
  A non-validated questionnaire that measures cooking attitudes and self-confidence will be used at baseline and after 8-months of follow-up. The "cooking self-confidence and attitudes questionnaire" includes 18 questions on self-confidence and 18 questions on attitudes. Each question includes a 5-item Likert scale answer. A higher score means a higher self-confidence or positive attitude on home cooking.

SECONDARY OUTCOMES:
Participants satisfaction | 3 months
  A non-validated "satisfaction questionnaire" will be used to identify potential barriers of the intervention, including time spent in each workshop with the chef and nutritionist, cost of the foods used in the workshops, and level of difficulty of the culinary techniques used in the study. Questions with a 5-item Likert scale answer will show a higher level of satisfaction with a higher score.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No